CLINICAL TRIAL: NCT05427656
Title: Imaging Biomarkers of Neuroplasticity and Neurodegeneration in the Living Human Brain (Uptake, Distribution and Pharmacokinetic) Study
Brief Title: Imaging Biomarkers of Neuroplasticity and Neurodegeneration in the Living Human Brain
Acronym: F18TRACK
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thiel, Alexander, M.D. (Individual)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MP-05-2023-3358
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Normal Healthy Adults

STUDY DESIGN:
Intervention Model Description: We will study a total of 30 participants, 10 in each of 3 age cohorts 18-29, 30-59 and 60-89, with equal numbers of male and female participants in each cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 185 MBq [18F] TRACK (Experimental): Each participant will receive a single scan with 185 MBq [18F] TRACK
  Interventions: Radiation: [18F] TRACK; Device: Measurement of Arterial Input Function

INTERVENTIONS:
Radiation: [18F] TRACK — We propose to use the radiotracer [18F] TRACK to non-invasively image the concentration of TrkB/C in the living human brain with PET in the 3 cohorts. The different subgroups of healthy controls will be used to define the best quantification method for our TrkB/C ligands and to assess a possible age dependency of TrkB/C binding in the healthy population, and may be of particular importance for the future study of patients with Alzheimer's Disease or mild cognitive impairment. Each participantsubject will receive a single scan with 185 MBq [18F] TRACK injected into an antecubital vein. Dynamic PET data will be acquired in list mode for 90 minutes ([18F] TRACK) respectively on a CTI/Siemens HRRT PET scanner at the brain imaging center of the Montreal Neurological Institute following our published procedure for [18F] TRACK after a transmission scan.
Device: Measurement of Arterial Input Function — The non-invasive detector, hereinafter called NID, comprises of plastic scintillating fibers (BCF-12, St-Gobain, France) wrapped in a medical-grade acrylic heat-shrink tube (Vention Medical, USA). The scintillating fibers are coupled to 5 m long transmission fibers to bring the signal out of the PET detector. The fibers will be held in place using a 3D-printed structure composed poly-lactic acid. The NID is designed to measure both positrons and photons escaping the wrist. Post-processing software is used to calculate the arterial input function.
  Other Names: Non-Invasive Detector

SUMMARY:
Following our recently completed whole body dosimetry study for [18F] TRACK in 6 healthy control subjects, the objective of this project is to evaluate brain uptake, regional distribution and in vivo pharmacokinetics for [18F] TRACK in 30 cognitively healthy controls using dynamic PET imaging. Specifically, we will evaluate [18F] TRACK in three cohorts of healthy control subjects of different ages and both sexes to further explore tracer kinetics in vivo and to determine the most appropriate and robust model to estimate tracer binding to TrkB/C. This will assess normal TrkB/C density in vivo and provide normative data for future use of these tracers in patients.

DETAILED DESCRIPTION:
We propose to use the radiotracer [18F] TRACK to non-invasively image the concentration of TrkB/C in the living human brain with Positron Emission Tomography in 3 different age cohorts. The different subgroups of healthy controls will be used to define the best quantification method for our TrkB/C ligands and to assess a possible age dependency of TrkB/C binding in the healthy population, that may be of particular importance for the future study of patients with Alzheimer's Disearse or mild cognitive impairment. We expect the proposed study to result in 1) a non-invasive method to quantify TrkB/C receptor binding in vivo, 2) age-specific norms of TrkB/C concentration and 3) a simplified approach for quantification which best approximates the full model without the need for arterial blood sampling for future use in patients.

ELIGIBILITY:
Inclusion Criteria:

In order to be considered a healthy control, participants will have a Clinical Dementia Rating (CDR) of 0, Montreal Cognitive Assessment (MoCA) greater than or equal to 26 and Mini-Mental State Exam (MMSE) of 24 or greater, with normal results on the Logical Memory 2 score from the Wechsler Memory Scale-Revise (cut-offs adjusted by education level), and normal scores on the Jessen questions for subjective memory complaints [21]. For the arterial catheter insertion, participants must have two viable arteries of the hand/arm. Women of childbearing potential must undergo a urine pregnancy test and may only be included if the urine pregnancy test is negative.

Exclusion Criteria:

Exclusion Criteria: When screening participants, we will question them as to whether they have participated in any other research studies over the past year in which they would have been exposed to radiation. Should they indicate that they have, we would not include them into the present study. A detailed questionnaire regarding Magnetic Resonance Imaging contraindications will be completed with each participant. Should they have any of the following, they will be excluded: cardiac pacemaker, an aneurysm clip, a metal prosthesis (e.g. artificial joints), an artificial heart valve or a metal clip on a blood vessel, metal in the eye or body, tattoos, body piercings, transdermal delivery systems (e.g. patch) or if they suffer from acute claustrophobia. Participants with any psychiatric or neurological conditions that could affect the brain will not be allowed to participate.

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Non-invasive method to quantify TrkB/C receptor binding in vivo | One Year
  Non-invasive method to quantify TrkB/C receptor binding in vivo
Age-specific norms of TrkB/C concentration | One Year
  Age-specific norms of TrkB/C concentration

SECONDARY OUTCOMES:
Arterial Input Function with Non-Invasive Detector | 2 months
  A simplified approach for quantification which best approximates the full model without the need for arterial blood sampling for future use in patients.

IPD SHARING:
Plan to Share IPD: No